CLINICAL TRIAL: NCT02919852
Title: Laparoscopic Retrovesical Colpopectinopexia in Treatment Pelvic Organ Prolapse
Brief Title: Laparoscopic Retrovesical Colpopectinopexia
Acronym: prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orel Regional Hospital, Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAV 31
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laparoscopic retrovesical colpopectinopexia (Other): new operative technic
  Interventions: Procedure: laparoscopic retrovesical colpopectinopexia

INTERVENTIONS:
Procedure: laparoscopic retrovesical colpopectinopexia — Laparoscopic correction of pelvic organ prolapse using a mesh in retrovesical space with pectineal ligament fixation.

SUMMARY:
The purpose of this study is to identify whether a new operative technic would be acceptable in female with pelvic organ prolapse.

DETAILED DESCRIPTION:
A new operative technic use to treat pelvic organ prolapse in women. Investigators plan to evaluate the results of procedure in the field of recurrence rate, effectiveness, mortality,morbidity and learning curves.

ELIGIBILITY:
Inclusion Criteria:

* all female with cystocele 1-2-3 grade? hysterocele 1-2 (POP-Q)

Exclusion Criteria:

* rectocele more then 1 grade (POP-Q) hysterocele more then 2

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
POP-Q assessment | first post operation day
  assessment of vaginal wall accordion to POP-Q score

SECONDARY OUTCOMES:
POP-Q assessment | 6 month after operation
  assessment of vaginal wall accordion to POP-Q score
POP-Q assessment | 1 year after operation
  assessment of vaginal wall accordion to POP-Q score

CONTACTS AND LOCATIONS:
Locations (1):
- LISOD, Kiev, Kyiv City, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided